CLINICAL TRIAL: NCT05077436
Title: A Randomised, Open-Label, Food Effect and Formulation Bioavailability Study of Two Vamifeport Oral Formulations in Healthy Male and Female Adults
Brief Title: Bioavailability Study Comparing 2 Vamifeport Oral Formulations in Fasted Versus Fed State in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vifor (International) Inc. (Industry)
Responsible Party: Sponsor
Organization: Vifor Pharma (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: VIT-2763-CP-103; 2021-003187-27 (EudraCT Number)
Record Dates: First submitted 2021-09-20; First posted 2021-10-14 (Actual); Last update posted 2022-08-17 (Actual); Status verified 2022-01

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Sequence 1 (Experimental): Participants receive a single dose of study drug, every 4 days:
  * Day 1: Participants in fasted state receive Vamifeport Formulation 1
  * Day 5: Participants in fed state receive Vamifeport Formulation 1
  * Day 9: Participants in fed state receive Vamifeport Formulation 2
  * Day 13: Participants in fasted state receive Vamifeport Formulation 2
  Interventions: Drug: Vamifeport Formulation 1; Drug: Vamifeport Formulation 2
- Sequence 2 (Experimental): Participants receive a single dose of study drug, every 4 days:
  * Day 1: Participants in fed state receive Vamifeport Formulation 1
  * Day 5: Participants in fasted state receive Vamifeport Formulation 2
  * Day 9: Participants in fasted state receive Vamifeport Formulation 1
  * Day 13: Participants in fed state receive Vamifeport Formulation 2
  Interventions: Drug: Vamifeport Formulation 1; Drug: Vamifeport Formulation 2
- Sequence 3 (Experimental): Participants receive a single dose of study drug, every 4 days:
  * Day 1: Participants in fasted state receive Vamifeport Formulation 2
  * Day 5: Participants in fed state receive Vamifeport Formulation 2
  * Day 9: Participants in fed state receive Vamifeport Formulation 1
  * Day 13: Participants in fasted state receive Vamifeport Formulation 1
  Interventions: Drug: Vamifeport Formulation 1; Drug: Vamifeport Formulation 2
- Sequence 4 (Experimental): Participants receive a single dose of study drug, every 4 days:
  * Day 1: Participants in fed state receive Vamifeport Formulation 2
  * Day 5: Participants in fasted state receive Vamifeport Formulation 1
  * Day 9: Participants in fasted state receive Vamifeport Formulation 2
  * Day 13: Participants in fed state receive Vamifeport Formulation 1
  Interventions: Drug: Vamifeport Formulation 1; Drug: Vamifeport Formulation 2

INTERVENTIONS:
Drug: Vamifeport Formulation 1 — Vamifeport Formulation 1 is available as 60 mg oral capsules
Drug: Vamifeport Formulation 2 — Vamifeport Formulation 2 is available as 60 mg oral capsules

SUMMARY:
Two different vamifeport oral formulations will be administered in fed and fasted state to assess the vamifeport food-drug interaction and to assess the relative bioavailability (the proportion of drug entering the circulation) of 2 different vamifeport oral formulations in healthy adult participants.

Participants will be randomly allocated to one of four treatment sequences, with four dosing periods each, where different combinations of both formulations will be administered following fasted and fed state.

The total study duration for each participant is up to 7 weeks and 4 days.

ELIGIBILITY:
Inclusion Criteria:

* Healthy participant. Healthy status defined by the Investigator.
* A body weight between 50 and 100 kg inclusive at screening.
* Non-smokers, or former smokers.
* Both female and male participants must agree to comply with the birth control requirements for the study.
* Ability to understand the requirements of the study and abide by the study restrictions, and agreement to return for the required assessments.

Exclusion Criteria:

* History of clinically significant gastrointestinal, cardiovascular, musculoskeletal, endocrine, neurological, hematological, psychiatric, renal, hepatic, bronchopulmonary, allergic or lipid metabolism disorders, cancer, or drug hypersensitivity.
* Any clinically relevant abnormal 12-lead ECG finding during screening or prior to randomization.
* A clinically relevant history of drug or alcohol misuse or abuse within 2 years prior to screening.
* Positive qualitative or semi-quantitative test for drugs of abuse positive cotinine screen (used to detect recent nicotine use), or alcohol breath test at screening (Visit 1) or Study Day -1 (Visit 2). Use of any of these agents will be not permitted during study participation.
* Strenuous physical exercise within the 1 week prior to Visit 2/Study Day -1 admission, and until completion of safety follow-up assessments are completed.
* Female participants who are pregnant or breastfeeding.
* Any concomitant medication (including herbal remedies and vitamins) taken within 2 weeks prior to Visit 2.
* Concomitant use of hormonal contraceptives (contraception associated with inhibition of ovulation), which are metabolized through cytochrome P450 (CYP) 3A4.
* Any other investigational drug.
* Blood draw or blood donation of ≥20 to <200 ml within 2 weeks, ≥200 to <400 ml within 4 weeks, or ≥400 ml within 12 weeks (male) or within 16 weeks (female) prior to Visit 2.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2021-10-14 (Actual); Primary Completion 2021-12-29 (Actual); Study Completion 2022-01-05 (Actual)

PRIMARY OUTCOMES:
Area under the plasma concentration versus time curve (AUC) from time 0 to the time of the last quantifiable concentration (AUC0-last) of vamifeport | Day 1, Day 5, Day 9, Day 13: 0-24 hours post-dose
Area under the plasma concentration versus time curve from time 0 extrapolated to infinite time (AUC0-infinity) of vamifeport | Day 1, Day 5, Day 9, Day 13: 0-24 hours post-dose
Maximum observed concentration (Cmax) of vamifeport | Day 1, Day 5, Day 9, Day 13: 0-24 hours post-dose

SECONDARY OUTCOMES:
Time of maximum vamifeport plasma concentration (Tmax) | Day 1, Day 5, Day 9, Day 13: 0-24 hours post-dose
Apparent terminal disposition phase half-life (tl/2) | Day 1, Day 5, Day 9, Day 13: 0-24 hours post-dose
Apparent terminal disposition phase rate constant | Day 1, Day 5, Day 9, Day 13: 0-24 hours post-dose
Apparent total clearance | Day 1, Day 5, Day 9, Day 13: 0-24 hours post-dose
Apparent volume of distribution during the terminal disposition phase | Day 1, Day 5, Day 9, Day 13: 0-24 hours post-dose

CONTACTS AND LOCATIONS:
Overall Officials: Peter Szecsödy, MD, Study Director — Clinical Research Director
Locations (1):
- Labcorp Clinical Research Unit Ltd., Leeds, United Kingdom

IPD SHARING:
Plan to Share IPD: No